CLINICAL TRIAL: NCT04027062
Title: Impact of Diabetes Continuing Education on Primary Health Care Physicians' Knowledge, Attitudes and Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Hosam Almetahr, Principal Investigator, King Khalid University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KingKalidU
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Diabete Mellitus
Keywords: Diabetes, Continuing education, Attitude, Practice, Health care physicians
MeSH Terms: conditions — Diabetes Mellitus; Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetes Continuing Education Program (Other): the physicians will be assessed before and after intervention
  the intervention group will be enrolled to the intervention program proposed to be (lecture + interactive workshop + group discussion + role play)
  Interventions: Behavioral: Diabetes Continuing Education Intervention

INTERVENTIONS:
Behavioral: Diabetes Continuing Education Intervention — The program will follow the International Curriculum for Diabetes Health Professional Education, which developed by the International Diabetes Federation (IFD) The key components of the proposed program content are Diabetes presentation and complications, Lifestyle, Nutrition, and Fitness.
  the intervention will be carried out by group of Diabetes educators from a different discipline, such as an Endocrinologist, Family physician, the dietitian will teach the attended physicians.

SUMMARY:
The main objective is to evaluate the effectiveness of a continuing education program on the Knowledge, Attitudes and Practices of primary health care physicians towards a high quality of diabetes care in Aseer region, Saudi Arabia.

DETAILED DESCRIPTION:
Background:

Diabetes is one of the rapidly growing chronic health conditions across the world. Healthcare providers still continue to face difficulties in delivering optimal care and education worldwide. Thus, continuing education is needed to improve Knowledge, Attitudes and Practices of physicians.

Objective: To evaluate the effectiveness of a continuing education (CE) program on the Knowledge, Attitudes and Practices of primary health care physicians (HCPs) towards a high quality of diabetes care.

Design and Methods:

This is a quasi-experimental design composed of pre-test post-test uncontrolled experimental design. The study will include all PHC physicians registered in health sectors of Abha and Khamis Musheet cities, Aseer Region. The physicians will be invited to attend a CE program. All participants will fill out a questionnaire before and after the intervention. The change in knowledge and attitudes of the participants will be measured at the end of the program. After 4 months, the practice of physicians will be assessed through retrospective review of patient's files.

Impact:

Education programs could positively influence the knowledge, beliefs and attitudes of healthcare workers toward a high quality of diabetes care, which in turn plays a major role in improving clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all PHC physicians registered in health sectors of Abha and Khamis musheet cities, Aseer Region
* willing to provide informed consent to participate in the study

Exclusion Criteria:

* physicians worked at hospital
* other health care professional (non-physicians)

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Percent of change of knowledge, attitude and practice of primary healthcare physicians | 4 months
  the primary outcome will be the difference between pre- and post-intervention regarding knowledge, attitude and practice of primary healthcare physicians.
  the knowledge and attitude will be assessed by questionnaire while the practice will be assessed through a retrospective review of patient's files.